CLINICAL TRIAL: NCT06832267
Title: A Single-center, Single-arm Phase II Trial of Rituximab-Methotrexate-Temozolomide-Thiotepa (RMTT) Regimen As First-line Therapy for Primary Central Nervous System Diffuse Large B-cell Lymphomas(PCNS DLBCL)
Brief Title: Rituximab-Methotrexate-Temozolomide-Thiotepa (RMTT) Regimen As First-line Therapy for PCNS DLBCL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang haiyan, Chief physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMTT
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Primary Central Nervous System Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rituximab-Methotrexate-Temozolomide-Thiotepa (RMTT) (Experimental): Rituximab: 375 mg/m2 intravenously on day 3,7; Methotrexate: 1.5-3.5 g/m2 intravenously on day 1,14(≤65 ,3.5g/m2；>65,1.5g/m2); Temozolomide 150 mg/m2 on days 3-7； Thiotepa:40 mg/m2 intravenously on day 17。 Treatment will be given for 4 cycles（28 days for each cycle）, and patients who achieve a CR or better can choose to undergo ASCT or WBRT(23.4Gy).
  Interventions: Drug: Rituximab-Methotrexate-Temozolomide-Thiotepa (RMTT)

INTERVENTIONS:
Drug: Rituximab-Methotrexate-Temozolomide-Thiotepa (RMTT) — Rituximab: 375 mg/m2 intravenously on day 3,7; Methotrexate: 1.5-3.5 g/m2 intravenously on day 1,14(≤65 ,3.5g/m2；>65,1.5g/m2); Temozolomide 150 mg/m2 on days 3-7； Thiotepa:40 mg/m2 intravenously on day 17。 Treatment will be given for 4 cycles（28 days for each cycle）, and patients who achieve a CR or better can choose to undergo ASCT or WBRT(23.4Gy).

SUMMARY:
This study aims to observe and explore the efficacy and safety of Rituximab-Methotrexate-Temozolomide-Thiotepa (RMTT) regimen as first-line therapy for primary central nervous system diffuse large B-cell lymphomas(PCNS DLBCL)

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily joined the study, signed the informed consent, and had good compliance;
* Patients with 18 Years to 75 Years(at the time of signing the informed consent); Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score: 0-3;
* Patients with histopathologically confirmed newly diagnosed primary central nervous system diffuse large B-cell lymphoma, and there were intracranial evaluable lesions (long diameter greater than 1.5cm, short diameter greater than 1cm);
* Patients who have not received any systemic therapy, except those who use hormones to control complications
* Expected survival of more than 3 months.
* Female patients of reproductive age should agree that birth control (such as intrauterine device, birth control pills, or condoms) must be used during the study period and for six months after completion; Having a negative serum pregnancy test within 7 days prior to study enrollment, and must be non-lactating; Male patients should agree to use contraception during the study period and for six months after the end of the study.

Exclusion Criteria:

* Patients who have previously received antitumor therapy or targeted therapy
* Patients who have undergone major surgery within the past 3 weeks .
* Presence of severe or uncontrolled comorbid conditions including, but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina, active peptic ulcer disease, or severe hemorrhagic disorders such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring transfusion or other medical interventions.
* Any active infection requiring systemic antimicrobial therapy within 14 days before starting study treatment, including, but not limited to, bacterial, fungal, and viral infections.
* Patients who are pregnant or breastfeeding.
* Current participation in other clinical studies, or initiation of study drugs administration less than 4 weeks after completion of previous clinical study treatment.
* Patients with concomitant diseases that, in the investigator's judgment, may seriously endanger patients' safety or may interfere with the completion of the study, or are deemed unsuitable for inclusion for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-02-14 (Estimated); Primary Completion 2027-02-13 (Estimated); Study Completion 2028-02-13 (Estimated)

PRIMARY OUTCOMES:
Complete Remission Rate（CRR） | Up to 16 weeks
  The proportion of subjects who achieves a best overall response of CR

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 16 weeks
  The proportion of subjects who achieves a best overall response of CR or PR.
Progression-Free Survival（PFS） | Up to 2 years
  From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first
overall survival(OS) | Up to 2 years
  The overall survival time refers to the time from therapy to death due to any cause.
Adverse event rate | From date of first day of treatment until 30 day after last treatment
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Yang, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No